CLINICAL TRIAL: NCT03542630
Title: Evaluation of Matrix Metalloproteinase 8 Salivary Test for Periodontal Diagnosis in Infertile Women
Brief Title: Evaluation of Matrix Metalloproteinase 8 Salivary Test for Diagnosis of Periodontitis
Status: Completed | Type: Observational
Sponsor: University of Zagreb (Other)
Responsible Party: Principal Investigator, Božana Lončar Brzak, Asisstant Professor, University of Zagreb
Other Study IDs: University of Zagreb
Record Dates: First submitted 2018-05-18; First posted 2018-05-31 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Periodontitis; Gingivitis; Infertility
MeSH Terms: conditions — Periodontitis; Gingivitis; Infertility | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — salivary samples for salivary MMP8 test
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- fertile, without periodontitis: Women who gave birth to at least one child, without preovious fertility treatments, and who do not have periodontitis.
  Interventions:
  salivary MMP8 test; periodontal examination; blood tests
  Interventions: Diagnostic Test: salivary MMP8 test; Other: periodontal examination; Other: blood tests
- fertile, with periodontitis: Women who gave birth to at least one child, without preovious fertility treatments, and who do have periodontitis.
  Interventions:
  salivary MMP8 test;periodontal examination;blood tests
  Interventions: Diagnostic Test: salivary MMP8 test; Other: periodontal examination; Other: blood tests
- infertile, without periodontitis: Women who are diagnosed with infertility of unknown cause, and who do not have periodontitis.
  Interventions:
  salivary MMP8 test; periodontal examination;blood tests
  Interventions: Diagnostic Test: salivary MMP8 test; Other: periodontal examination; Other: blood tests
- infertile, with periodontitis: Women who are diagnosed with infertility of unknown cause, and who do have periodontitis.
  Interventions:
  salivary MMP8 test; periodontal examination; blood tests
  Interventions: Diagnostic Test: salivary MMP8 test; Other: periodontal examination; Other: blood tests

INTERVENTIONS:
Diagnostic Test: salivary MMP8 test — All female participants will make salivary MMP8 test and certain blood parameters to determine systemic inflammatory response
Other: periodontal examination — Periodontal examination by a specialist of periodontology will be made to all female participants, using periodontal probe and dental mirror.
Other: blood tests — All female participants who do not have recent blood tests will make new blood tests to determine certain blood parameters.

SUMMARY:
Despite the great progress in understanding the causes of infertility, the reason for the failure of pregnancy has not been discovered among 25% of infertile couples. Some studies have shown the negative impact of periodontal disease on the reproductive potential of women. It is known that there is an elevated level of matrix metalloproteinase 8 (MMP8) in the gingival fluid of patients with periodontitis. It is possible to establish a fast diagnosis of periodontitis by using a non-invasive assay based on monoclonal antibodies to two epitopes of MMP-8. The goal of the research is to use the above described assay in order to compare the level of MMP8 in the gingival fluid of infertile patients with the control group of fertile women, depending on the existence of periodontal disease. It is expected to find significantly higher values of MMP8 in infertile patients in relation to the fertile patient with/without periodontitis. The prompt treatment of periodontitis in preconception care of this group of women could have a significant impact on the improvement of fertility and ability to achieve pregnancy.

DETAILED DESCRIPTION:
Periodontal disease or periodontitis is a common chronic infection and inflammatory gingival disease and its supportive tissue associated with several unwanted effects, including serious obstetric consequences. Periodontitis is commonly diagnosed in clinical practice based on clinical findings and radiological examinations, but also with the help of microbiological or periodontal bacterial specimens. Several salivary markers have been investigated and it appears that the determination of matrix metalloproteinases provides clear information on the difference between gingivitis, periodontitis, and healthy periodontitis. Especially in this respect, matrix metalloproteinase 8 (MMP 8) was investigated, which proved to be a fairly good marker. Little is known about the effect of periodontitis on reproductive potential of women. Some studies have assumed that periodontitis could be one of the possible risk factors of infertility of an unknown cause. One of the possible mechanisms responsible for the negative influence of periodontitis is the conception of the mediator of inflammation at the level of the endometrium and the place of implantation of the embryo.The aim of the study was to compare the level of MMP8 in salivary fluid in infertile patients in relation to the control group of fertile women, depending on the existence of periodontitis.

ELIGIBILITY:
Inclusion Criteria:

* fertile women- women who gave birth to at least one child, without previous fertility treatments, with or without periodontitis
* infertile women- women who are diagnosed with infertility of unknown cause, with or without periodontitis

Exclusion Criteria:

* female with known cause of infertility

Ages: 25 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: The study will comprise a total of 100 women, of which 25 fertile women without periodontitis; 25 fertile women, with periodontitis; 25 infertile women, with unknown cause of infertility and with periodontitis and 25 infertile women with unknown cause of infertility and without periodontitis.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Salivary MMP8 test for diagnostics of periodontitis | 2018-2019
  Evaluation of salivary MMP8 test for diagnostics of periodontitis

CONTACTS AND LOCATIONS:
Overall Officials: Božana Lončar Brzak, Assist.Prof., Principal Investigator — University of Zagreb
Locations (1):
- School of Dental Medicine, University of Zagreb, Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mantyla P, Stenman M, Kinane DF, Tikanoja S, Luoto H, Salo T, Sorsa T. Gingival crevicular fluid collagenase-2 (MMP-8) test stick for chair-side monitoring of periodontitis. J Periodontal Res. 2003 Aug;38(4):436-9. doi: 10.1034/j.1600-0765.2003.00677.x. PMID 12828663
- [Background] Hart R, Doherty DA, Pennell CE, Newnham IA, Newnham JP. Periodontal disease: a potential modifiable risk factor limiting conception. Hum Reprod. 2012 May;27(5):1332-42. doi: 10.1093/humrep/des034. Epub 2012 Feb 22. PMID 22362927
- [Background] Kraft-Neumarker M, Lorenz K, Koch R, Hoffmann T, Mantyla P, Sorsa T, Netuschil L. Full-mouth profile of active MMP-8 in periodontitis patients. J Periodontal Res. 2012 Feb;47(1):121-8. doi: 10.1111/j.1600-0765.2011.01416.x. Epub 2011 Sep 30. PMID 21958332
- See also: related information — https://www.ncbi.nlm.nih.gov/pubmed/?term=Hart+R%2C+Doherty+DA%2C+Pennell+CE%2C+Newnham+IA%2C+Newnham+JP.+Periodontal+disease%3A+a+potential+modifiable+risk+factor+limiting+conception.